CLINICAL TRIAL: NCT04694859
Title: Romanian National Registry of Outcomes After Transcatheter Aortic Valve Implantation in Patients With Severe Aortic Stenosis - RO-TAVI
Acronym: RO-TAVI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Romanian Society of Cardiology (Other)
Responsible Party: Sponsor
Other Study IDs: RO-TAVI
Record Dates: First submitted 2020-12-31; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Aortic Stenosis Symptomatic; Aortic Valve Stenosis
Keywords: aortic stenosis
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Symptomatic Severe Aortic Valve Stenosis: Patients >18 years old with symptomatic severe aortic valve stenosis.
  Interventions: Device: Transcatheter Aortic Valve Implantation

INTERVENTIONS:
Device: Transcatheter Aortic Valve Implantation — Transfemoral or transapical Transcatheter Aortic Valve Implantation

SUMMARY:
RO-TAVI is a national prospective, observational, multi-center registry registry of patients with aortic valve stenosis undergoing transcatheter aortic valve implantation (TAVI) to assess patient care and outcomes.

DETAILED DESCRIPTION:
Background: Since the establishment of transcatheter aortic valve implantation (TAVI) in Romania in 2015 there has been a growing number of interventions being performed by an increasing number of hospitals throughout the country. In 2018, there were more than 250 implants, which are expected to grow in the following years by about 30% on an annual basis.

Objective: This is a national quality assurance initiative to improve patient care and outcomes. It further serves as a database for the assessment of the safety and efficacy of TAVI and its financial implications (e.g. reimbursement).

Design: National, prospective, observational, multi-center registry. All centers performing TAVI in Romania; minimum cases per center for inclusion: 20 cases/year-to-date Population: All patients undergoing TAVI in Romania at any of the participating centers with a CE-marked valve of any manufacturer given that they provide written informed consent.

ELIGIBILITY:
Inclusion Criteria:

* severe symptomatic aortic valve stenosis
* high risk or patients deemed amenable for TAVI by a multidisciplinary team
* signed informed consent to participate in the study

Exclusion Criteria:

* inadequate annulus size (<18 mm, >29 mm)
* left ventricle thrombus
* active endocarditis
* high risk of coronary ostium obstruction
* plaques with mobile thrombi in the ascending aorta, or arch
* hemodynamic instability
* estimated life expectancy <1 year
* comorbidity suggesting lack of improvement of quality of life
* other situations adjudicated by the local HeartTeam

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years old diagnosed with symptomatic severe aortic valve stenosis undergoing TAVI.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-01-05 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Mortality | 1-year
  All cause mortality

SECONDARY OUTCOMES:
Stroke | 1-year
  Ischemic or hemorrhagic cerebrovascular accident
Bleeding | 1-year
  Major bleeding
Myocardial ischemia | 1-year
  Acute myocardial infarction or recurrent angina
Arrhythmia | 1-year
  Arrhythmias requiring permanent pacemaker implantation
Vascular complications | 1-year
  Procedure related vascular complications
Acute kidney injury | 1-year
  Procedure related renal dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Vlad A Iliescu, MD PhD, Principal Investigator — University of Medicine and Pharmacy "Carol Davila", Bucharest, Romania; Bogdan A Popescu, MD PhD, Principal Investigator — University of Medicine and Pharmacy "Carol Davila", Bucharest, Romania; Dragos Vinereanu, MD PhD, Principal Investigator — University of Medicine and Pharmacy "Carol Davila", Bucharest, Romania
Locations (1):
- Catalina A. Parasca, MD, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lindroos M, Kupari M, Heikkila J, Tilvis R. Prevalence of aortic valve abnormalities in the elderly: an echocardiographic study of a random population sample. J Am Coll Cardiol. 1993 Apr;21(5):1220-5. doi: 10.1016/0735-1097(93)90249-z. PMID 8459080
- [Background] Vahanian A, Alfieri O, Andreotti F, Antunes MJ, Baron-Esquivias G, Baumgartner H, Borger MA, Carrel TP, De Bonis M, Evangelista A, Falk V, Lung B, Lancellotti P, Pierard L, Price S, Schafers HJ, Schuler G, Stepinska J, Swedberg K, Takkenberg J, Von Oppell UO, Windecker S, Zamorano JL, Zembala M; ESC Committee for Practice Guidelines (CPG); Joint Task Force on the Management of Valvular Heart Disease of the European Society of Cardiology (ESC); European Association for Cardio-Thoracic Surgery (EACTS). Guidelines on the management of valvular heart disease (version 2012): the Joint Task Force on the Management of Valvular Heart Disease of the European Society of Cardiology (ESC) and the European Association for Cardio-Thoracic Surgery (EACTS). Eur J Cardiothorac Surg. 2012 Oct;42(4):S1-44. doi: 10.1093/ejcts/ezs455. Epub 2012 Aug 25. No abstract available. PMID 22922698
- [Background] Kodali SK, Williams MR, Smith CR, Svensson LG, Webb JG, Makkar RR, Fontana GP, Dewey TM, Thourani VH, Pichard AD, Fischbein M, Szeto WY, Lim S, Greason KL, Teirstein PS, Malaisrie SC, Douglas PS, Hahn RT, Whisenant B, Zajarias A, Wang D, Akin JJ, Anderson WN, Leon MB; PARTNER Trial Investigators. Two-year outcomes after transcatheter or surgical aortic-valve replacement. N Engl J Med. 2012 May 3;366(18):1686-95. doi: 10.1056/NEJMoa1200384. Epub 2012 Mar 26. PMID 22443479
- [Background] Kappetein AP, Head SJ, Genereux P, Piazza N, van Mieghem NM, Blackstone EH, Brott TG, Cohen DJ, Cutlip DE, van Es GA, Hahn RT, Kirtane AJ, Krucoff MW, Kodali S, Mack MJ, Mehran R, Rodes-Cabau J, Vranckx P, Webb JG, Windecker S, Serruys PW, Leon MB; Valve Academic Research Consortium (VARC)-2. Updated standardized endpoint definitions for transcatheter aortic valve implantation: the Valve Academic Research Consortium-2 consensus document (VARC-2). Eur J Cardiothorac Surg. 2012 Nov;42(5):S45-60. doi: 10.1093/ejcts/ezs533. Epub 2012 Oct 1. PMID 23026738
- [Background] Iung B, Delgado V, Rosenhek R, Price S, Prendergast B, Wendler O, De Bonis M, Tribouilloy C, Evangelista A, Bogachev-Prokophiev A, Apor A, Ince H, Laroche C, Popescu BA, Pierard L, Haude M, Hindricks G, Ruschitzka F, Windecker S, Bax JJ, Maggioni A, Vahanian A; EORP VHD II Investigators. Contemporary Presentation and Management of Valvular Heart Disease: The EURObservational Research Programme Valvular Heart Disease II Survey. Circulation. 2019 Oct;140(14):1156-1169. doi: 10.1161/CIRCULATIONAHA.119.041080. Epub 2019 Sep 12. PMID 31510787